CLINICAL TRIAL: NCT05520736
Title: Implementing a Mobile Health Supported Bundle to Improve Routine Vaccination Completion Rate in a Low-resource Setting
Brief Title: Mhealth Supported Bundle to Improve Vaccination Completion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Osayame Ekhaguere, Assistant Professor, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 15107; KL2TR002530 (NIH); UL1TR002529 (NIH)
Record Dates: First submitted 2022-08-26; First posted 2022-08-30 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Vaccination
Keywords: Vaccination; Childhood; Low- and middle-income country
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Prospectively received appointment reminders, motivational interviews and targeted vaccine drives.
  Interventions: Behavioral: Appointment reminders, motivational interviewing and targeted vaccine drives

INTERVENTIONS:
Behavioral: Appointment reminders, motivational interviewing and targeted vaccine drives — Automated and real time phone call reminders, motivational interviewing and targeted vaccine drives applied in sequence

SUMMARY:
Supported be a digital vaccine registry the investigators will test the impact of automated appointment reminders, real time appointment reminders, motivational interviewing and targeted vaccine on routine childhood vaccine completion rates.

DETAILED DESCRIPTION:
Bundling three high-impact mHealth interventions (a digital vaccine registry (supply side), a reminder system (demand side), and targeted vaccine drive (demand and supply-side) will be feasible, acceptable, carried out with fidelity, and result in a 10% improvement in vaccine completion rates compared to the year prior to implementation.

ELIGIBILITY:
Inclusion Criteria:

* All parents or caregivers of patients who bring their child to the vaccine clinic to receive immunization for their first vaccine visit.

Exclusion Criteria:

* Parents or caregivers not willing to participate.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2855 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
DPT3 vaccine completion rate | 15 Months
  The proportion of enrolled subjects who complete the Diphtheria, pertussis, and tetanus vaccine (DPT3) vaccine series when assessed at 15 months of age.
Measles vaccine completion rate | 15 Months
  The proportion of enrolled subjects who complete the measles vaccine series when assessed at 15 months of age.
Number of eligible subjects enrolled | 15 Months
  Vaccine clinic records will be reviewed to identify the total number of eligible patients in the clinic (defined as those presenting to the vaccine clinic with a child receiving their first vaccine) and the number who agreed to participate during the study period.
Provider Adoption | 15 Months
  A modified intervention acceptability, perception and system usability assessment using a Likert scale questionnaire.
Protocol Adherence | 15 Months
  The proportion of eligible subjects who received a real-time phone call reminder, counselling, and targeted vaccine drive when indicated
Project Cost | 15 Months
  The cost of administering each component of the mHealth bundle will be documented, such as cost of targeted drive and cost of real time phone calls. This will assist in determining the cost to scale the project.

CONTACTS AND LOCATIONS:
Overall Officials: Osayame A Ekhaguere, Principal Investigator — Indiana University
Locations (1):
- Mother and Child Hospital Akure, Akure, Ondo State, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
Publish a study protocol in an open access journal. Provider study data set on request.
Supporting Information: Study Protocol, CSR
Time Frame: Protocol: Within 6 month of study start Data set: After study completion.
Access Criteria: One request